CLINICAL TRIAL: NCT02299869
Title: Comparative Study to Evaluate the Cosmetic Appearance of Two Brands (Coopervision (CVI) vs. Competitor) of Color Soft Contact Lenses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EX-MKTG-51
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 - Verde (Competitor-control) vs. Green (CVI-test) (Other): Each subject was randomized to wear the test and control lenses contralaterally.
  Interventions: Device: Verde (Competitor-control); Device: Green (CVI-test)
- Group 2 - Cinza (Competitor-control) vs. Grey (CVI-test) (Other): Each subject was randomized to wear the test and control lenses contralaterally.
  Interventions: Device: Cinza (Competitor-control); Device: Grey (CVI-test)
- Group 3 - Esmeralda (Competitor-control) vs. Jade (CVI-test) (Other): Each subject was randomized to wear the test and control lenses contralaterally.
  Interventions: Device: Esmeralda (Competitor-control); Device: Jade (CVI-test)
- Group 4 - Azul (Competitor-control) vs. Blue (CVI-test) (Other): Each subject was randomized to wear the test and control lenses contralaterally.
  Interventions: Device: Azul (Competitor-control); Device: Blue (CVI-test)

INTERVENTIONS:
Device: Verde (Competitor-control) — contact lens
  Other Names: methafilcon A
  Arms: Group 1 - Verde (Competitor-control) vs. Green (CVI-test)
Device: Green (CVI-test) — contact lens
  Other Names: methafilcon A
  Arms: Group 1 - Verde (Competitor-control) vs. Green (CVI-test)
Device: Cinza (Competitor-control) — contact lens
  Other Names: methafilcon A
  Arms: Group 2 - Cinza (Competitor-control) vs. Grey (CVI-test)
Device: Grey (CVI-test) — contact lens
  Other Names: methafilcon A
  Arms: Group 2 - Cinza (Competitor-control) vs. Grey (CVI-test)
Device: Esmeralda (Competitor-control) — contact lens
  Other Names: methafilcon A
  Arms: Group 3 - Esmeralda (Competitor-control) vs. Jade (CVI-test)
Device: Jade (CVI-test) — contact lens
  Other Names: methafilcon A
  Arms: Group 3 - Esmeralda (Competitor-control) vs. Jade (CVI-test)
Device: Azul (Competitor-control) — contact lens
  Other Names: methafilcon A
  Arms: Group 4 - Azul (Competitor-control) vs. Blue (CVI-test)
Device: Blue (CVI-test) — contact lens
  Other Names: methafilcon A
  Arms: Group 4 - Azul (Competitor-control) vs. Blue (CVI-test)

SUMMARY:
Comparative Study to Evaluate the Cosmetic Appearance of Two Brands (Coopervision (CVI) vs. Competitor)of Color Soft Contact Lenses

DETAILED DESCRIPTION:
Each lens pair comparison will require two visits over two days, as follows: Visits: V1 (lens dispensing), V2 (20 minutes post lens settling). Each subject will be randomized to wear the test and control lenses in a series of four short fitting comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive).
* Has had a self-reported visual exam in the last two years.
* Is an adapted wearer of spherical soft contact lenses.
* Has a contact lens spherical prescription between - 1.00 and - 10.00 (inclusive).
* Has a spectacle cylinder up to 0.75 diopter (D) in each eye
* Can achieve best corrected spectacle distance visual acuity of 20/30 (0.18 logMAR) or better in each eye.
* Has clear corneas and no active ocular disease.
* Has read, understood and signed the information consent letter.
* Is willing to wear his/hers spectacles over the study contact lenses.
* Is willing to comply with the wear schedule.
* Is willing to comply with the visit schedule.

Exclusion Criteria:

* Has never worn contact lenses before.
* Currently wears rigid gas permeable contact lenses.
* Has a history of not achieving comfortable contact lens wear (5 days per week; > 8 hours/day)
* Has a contact lens prescription outside the range of - 1.00 to -10.00D.
* Has a spectacle cylinder ≥1.00D of cylinder in either eye.
* Does not have a pair of corrective spectacles at the time of the visit.
* Cannot achieve best corrected spectacle distance visual acuity of 20/30 (0.18 logMAR) or better in each eye.
* Presence of clinically significant (grade > 2.0, scale 0-4) anterior segment abnormalities.
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (past or present)
  * Seborrheic eczema, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-10; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Velazquez Guerrero, MSc FIACLE, Principal Investigator — School of Optometry, National Autonomous University (UNAM), Mexico
Locations (1):
- Optometry Clinic, National Autonomous University, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was disqualified from the study due to not meeting inclusion criteria before lens dispensing.
Period: Overall Study
Arm/Group | Group 1 - Verde (Competitor-control) vs. Green (CVI-test) | Group 2 - Cinza (Competitor-control) vs. Grey (CVI-test) | Group 3 - Esmeralda (Competitor-control) vs. Jade (CVI-test) | Group 4 - Azul (Competitor-control) vs. Blue (CVI-test)
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Verde (Competitor-control) vs. Green (CVI-test) | Group 2 - Cinza (Competitor-control) vs. Grey (CVI-test) | Group 3 - Esmeralda (Competitor-control) vs. Jade (CVI-test) | Group 4 - Azul (Competitor-control) vs. Blue (CVI-test) | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.5 (2.3) | 21.8 (2.3) | 20.7 (2.4) | 20.9 (1.9) | 21.2 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 10 | 9 | 33
  Male | 1 | 5 | 0 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Cosmetic Appearance Preference
Description: Participant's subjective preference for cosmetic appearance. 3 point Likert Scale. 1=prefer CVI-test lens 2=prefer Competitor-control lens, 3=no preference
Time Frame: 20 minutes
Measure: Number; unit: participants
Arm/Group | Group 1 - Verde (Competitor-control) vs. Green (CVI-test) | Group 2 - Cinza (Competitor-control) vs. Grey (CVI-test) | Group 3 - Esmeralda (Competitor-control) vs. Jade (CVI-test) | Group 4 - Azul (Competitor-control) vs. Blue (CVI-test)
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants
  Competitor-control lens | 8 | 9 | 4 | 5
  CVI-test lens | 2 | 1 | 5 | 4
  No preference | 0 | 0 | 1 | 1

2. Primary Outcome: Comfort
Description: Participant's subjective rating for comfort. (Scale 0-10, 0=poor, 10=excellent).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 - Verde (Competitor-control) vs. Green (CVI-test) | Group 2 - Cinza (Competitor-control) vs. Grey (CVI-test) | Group 3 - Esmeralda (Competitor-control) vs. Jade (CVI-test) | Group 4 - Azul (Competitor-control) vs. Blue (CVI-test)
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Competitor-control lens | 8.6 (2.2) | 7.1 (2.3) | 8.2 (1.7) | 7.1 (2.2)
  CVI-test lens | 7.3 (1.7) | 8.2 (1.9) | 7.0 (2.9) | 8.0 (2.1)

3. Primary Outcome: Comfort
Description: Participant's subjective rating for comfort. (Scale 0-10, 0=poor, 10=excellent).
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 - Verde (Competitor-control) vs. Green (CVI-test) | Group 2 - Cinza (Competitor-control) vs. Grey (CVI-test) | Group 3 - Esmeralda (Competitor-control) vs. Jade (CVI-test) | Group 4 - Azul (Competitor-control) vs. Blue (CVI-test)
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale
  Competitor control lens | 9.3 (0.8) | 8.3 (1.2) | 8.6 (1.0) | 8.1 (1.8)
  CVI-test lens | 7.5 (1.7) | 8.0 (1.9) | 7.3 (2.0) | 8.8 (1.4)

4. Primary Outcome: Comfort Preference
Description: Participant's subjective preference for comfort on a 3 point Likert Scale. 1=prefer CVI-test lens, 2=prefer Competitor-control lens, 3=no preference
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Group 1 - Verde (Competitor-control) vs. Green (CVI-test) | Group 2 - Cinza (Competitor-control) vs. Grey (CVI-test) | Group 3 - Esmeralda (Competitor-control) vs. Jade (CVI-test) | Group 4 - Azul (Competitor-control) vs. Blue (CVI-test)
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants
  Competitor-control lens | 9 | 4 | 3 | 3
  CVI-test lens | 1 | 4 | 5 | 6
  No preference | 0 | 2 | 2 | 1

5. Primary Outcome: Comfort Preference
Description: as for outcome 4
Time Frame: 20 minutes
Measure: Number; unit: participants
Arm/Group | Group 1 - Verde (Competitor-control) vs. Green (CVI-test) | Group 2 - Cinza (Competitor-control) vs. Grey (CVI-test) | Group 3 - Esmeralda (Competitor-control) vs. Jade (CVI-test) | Group 4 - Azul (Competitor-control) vs. Blue (CVI-test)
Number analyzed (Participants) | 10 | 10 | 10 | 10
participants
  Competitor-control lens | 8 | 4 | 4 | 4
  CVI-test lens | 2 | 6 | 5 | 4
  No preference | 0 | 0 | 1 | 2

ADVERSE EVENTS:
Groups:
- Overall Participants: Each subject was randomized to wear the test and control lenses in a series of four short fitting comparisons (pair 1, pair 2, pair 3, and pair 4).
Arm/Group | Overall Participants
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other